CLINICAL TRIAL: NCT06741774
Title: Efficacy and Safety of Trabecular Meshwork Microstent Drainage System in Reducing Intraocular Pressure in Adult Patients with Mild to Moderate Open-angle Glaucoma Combined with Cataract: a Prospective, Multicenter, Randomized, Open Label, Parallel Controlled, Superiority Clinical Trial
Brief Title: Efficacy and Safety of Trabecular Meshwork Microstent Drainage System ( MicroCOGO )
Acronym: MicroCOGO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Healthguard Biomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGB-CMP-TMS-001
Record Dates: First submitted 2024-12-09; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Open-angle Glaucoma; Cataract
Keywords: cataract; IOP reduction; open-angle glaucoma; trabecular meshwork; micro stent
MeSH Terms: conditions — Glaucoma, Open-Angle; Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- combined phacoemulsification and implantation of Trabecular Meshwork Microstent Drainage System (Experimental): Eyes with OAG and cataracts randomly divided into test group that were planned for combined phacoemulsification and implantation of Trabecular Meshwork Microstent Drainage System.
  Interventions: Device: Trabecular Meshwork Microstent Drainage System
- phacoemulsification (Active Comparator): Eyes with OAG and cataracts randomly divided into control group that were planned for phacoemulsification alone.
  Interventions: Procedure: phacoemulsification

INTERVENTIONS:
Device: Trabecular Meshwork Microstent Drainage System — The device is implanted on the functional trabecular meshwork with head in schlemm canal and tail in anterior chamber. There is a hollow tube connecting schlemm canal and anterior chamber. The device can promote external drainage of aqueous humor to reduce intraocular pressure.
  Other Names: combined phacoemulsification and implantation of Trabecular Meshwork Microstent Drainage System
  Arms: combined phacoemulsification and implantation of Trabecular Meshwork Microstent Drainage System
Procedure: phacoemulsification — Eyes with OAG and cataracts randomly divided into control group that were planned for phacoemulsification alone.
  Arms: phacoemulsification

SUMMARY:
It is a prospective, multicenter, randomized, open label, parallel controlled, superiority clinical trial that evaluate efficacy and safety of Trabecular Meshwork Microstent Drainage System in Reducing Intraocular Pressure in Adult Patients With Mild to Moderate Open-angle Glaucoma Combined With Cataract.

DETAILED DESCRIPTION:
The trial is a prospective, multicenter, randomized, open label, parallel controlled, superiority study. Eligible subjects will be randomly assigned to either test group or control group for treatment. The trial is divided into four research stages, with each subject expected to participate for maximum 14 months. The entire research phase includes:

Screening visit (V1, -60~-1 day). Baseline visit (V2). Randomization and surgery (V3): The subjects will be randomly assigned in 2:1 ratio to either test group (phacoemulsification with implantation of IOL combined with implantation of trabecular meshwork microstent drainage system) or control group (phacoemulsification with implantation of IOL only).

Follow-up visits (V4 ~ V10): different time points after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male of female, age 18 years or older
* Mild to moderate open-angle glaucoma
* Cataract
* Average of IOP is less than or equal to 24mmHg with 1-3 drugs in the screening period
* All 3 diurnal IOPs after drug-eluting are greater than 21mmHg and less than or equal to 35mmHg, average of diurnal IOPs is at least 3.0mmHg higher than the pre drug-eluting IOP
* Cup to disc ratio (C/D) less than or equal to 0.8, or VFI greater than 75%
* Gonioscope shows that anterior chamber angle is open

Exclusion Criteria:

* Traumatic, uveitic, neovascular, angle-closure glaucoma or glaucoma associated with vascular disorders
* Active corneal inflammation or edema
* Retinal disorders not associated with glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2025-12-04 (Estimated); Study Completion 2026-05-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with reduction of IOP greater than or equal to 20% compared to baseline in 12th month after surgery | 12 months
  IOP measured by Goldmann applanation tonometry

CONTACTS AND LOCATIONS:
Overall Officials: Xinghuai Sun, Doctor, Principal Investigator — EENT hospital of Fudan University
Locations (1):
- Healthguard Biomed, Suzhou, Jiangsu, China